CLINICAL TRIAL: NCT02250404
Title: Pilot Study of the Identification of the Molecular Signatures of Relapse in Small Cell Lung Cancer
Brief Title: Molecular Signatures of Relapse in Tissue Samples From Patients With Small Cell Lung Cancer Who Are Receiving Cisplatin and Etoposide
Status: Withdrawn | Type: Observational
Why Stopped: PI left institution
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2O-13-1; NCI-2014-01910 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HS-14-00382; 2O-13-1 (Other: USC Norris Comprehensive Cancer Center); UL1TR000130 (NIH); P30CA014089 (NIH)
Record Dates: First submitted 2014-09-23; First posted 2014-09-26 (Estimated); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (molecular profile): Previously collected tissue samples are analyzed via RNA sequencing and DNA methylation at baseline. Patients also undergo collection of tissue samples for analysis at relapse.
  Interventions: Other: cytology specimen collection procedure; Other: laboratory biomarker analysis

INTERVENTIONS:
Other: cytology specimen collection procedure — Correlative studies
  Other Names: cytologic sampling
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This pilot research trial studies molecular signatures of the return of cancer after a period of improvement (relapse) in tissue samples from patients with small cell lung cancer who are receiving or planning to receive cisplatin and etoposide. Studying samples of tissue from patients with small cell lung cancer in the laboratory may help doctors learn more about the changes that occur in deoxyribonucleic acid (DNA) and identify biomarkers related to cancer relapse.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To collect and analyze small cell lung cancer (SCLC) tumor DNA and ribonucleic acid (RNA) from 3 human patients before and after relapse to identify the molecular signatures of relapse.

OUTLINE:

Previously collected tissue samples are analyzed via RNA sequencing and DNA methylation at baseline. Patients also undergo collection of tissue samples for analysis at relapse.

ELIGIBILITY:
Inclusion Criteria:

* Any patient seen at Norris or County with histologically confirmed SCLC, with tissue in the Norris Cancer Center Tumor Repository
* Patients must be undergoing or about to start first line treatment with cisplatin and etoposide
* Patients may not have a second malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects seen at USC Norris Comprehensive Cancer Center and at LAC USC Medical Center with histologically confirmed small cell lung cancer will be recruited for this trial.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-08-22 (Actual); Primary Completion 2018-08-22 (Estimated); Study Completion 2019-08-22 (Estimated)

PRIMARY OUTCOMES:
Change in tumor tissue molecular profiles | Baseline to up to 1 year
  Profiles of pre- and post-relapse tumor tissue will be compared. Data will be compared with mouse data and overlaps determined.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Gitlitz, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California